CLINICAL TRIAL: NCT03456661
Title: Comparison Between Levobupivacaine 0.25% and Levobupivacaine With Dexmedetomidine in Ultrasound Guided Modified Pectoral Nerve Block, a Double Blind Randomised Controlled Trial.
Brief Title: Comparison Between Levobupivacaine and Levobupivacaine With Dexmedetomidine in Ultrasound Guided Pectoral Nerve Block
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The surgical approach has changed.
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Hilde Coppejans, data manager, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2014-002589-56; B300201421166 (Registry Identifier: FAGG)
Record Dates: First submitted 2014-08-08; First posted 2018-03-07 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer; Mastectomy, Modified Radical
Keywords: Pectoral block; Ultrasound; Mastectomy; Levobupivacaine; Dexmedetomidine
MeSH Terms: conditions — Breast Neoplasms | interventions — Levobupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levobupivacaine (Active Comparator): Study Group 1 (Group L): patients undergoing an ultrasound guided modified pectoral nerve block (technique described by Blanco et al[1]) with levobupivacaine 0.25% 29,5ml + 0,5ml physiologic serum (total volume 30ml) (10ml between major and minor pectoral muscle and 20ml between minor pectoral muscle and anterior serratus muscle at the level of the third or fourth rib).
  Interventions: Drug: Levobupivacaine
- Levobupivacaine + Dexmedetomidine (Active Comparator): Study Group 2 (Group LD): patients undergoing an ultrasound guided modified pectoral nerve block (a technique described by Blanco et al[1]) with levobupivacaine 0.25% 29,5ml + Dexmedetomidine 50µg (0,5ml)with a total volume of 30ml. (10ml between major and minor pectoral muscle and 20ml between minor pectoral muscle and anterior serratus muscle at the level of the third or fourth rib).
  Interventions: Drug: Levobupivacaine + Dexmedetomidine

INTERVENTIONS:
Drug: Levobupivacaine — Infiltration with 0.25% 29,5ml + 0,5ml physiologic serum (total volume 30ml), US guided, using pectoralis block technique.
  Other Names: Chirocaine
  Arms: Levobupivacaine
Drug: Levobupivacaine + Dexmedetomidine — Infiltration with chirocaine 0.25% 29,5ml + 0,5ml dexmedetomidine (50µg) (total volume 30ml), US guided, using pectoralis block technique.
  Arms: Levobupivacaine + Dexmedetomidine

SUMMARY:
A double blind prospective randomized controlled trial in which the effect of single shot levobupivacaine 0,25% will be compared with the effect of levobupivacaine 0.25% in association with dexmedetomidine when performing an ultrasound guided modified pectoral nerve block , in patients undergoing a mastectomy with axillar procedure.

The difference in effect will be evaluated by monitoring the postoperative morphine consumption in both groups .

The hypothesis is that there is a significant decrease in morphine consumption during the first 24h postoperatively due to association of dexmedetomidine to the local anesthetic compared to the local anesthetic alone when performing a ultrasound guided modified pectoral nerve block. The morphine consumption will be the primary outcome parameter.

DETAILED DESCRIPTION:
Women (18+, American Society of Anesthesiologists 1,2,3) undergoing a mastectomy with axillar procedure will be randomised and receive a ultrasound guided modified pectoral nerve block, if participants meet in- and exclusion criteria and provide written informed consent.

Using a two needle approach, ten milliliters of local anesthetic is injected under ultrasound guidance between the major and minor pectoral muscle and twenty milliliters between the minor pectoral and the serratus anterior muscle, on the side to be operated.

Participants receive intravenous Patient Controlled Analgesia with morphine and dehydrobenzperidol (1mg/ml morphine, 50µg dehydrobenzperidol/ml).

Furthermore every participant in the trial will receive ketorolac 0.5mg/kg three times a day and paracetamol four times 1g per day.

When the analgesia using the intravenous Patient Controlled Analgesia regime isn't sufficient, the anesthesiologist will titrate with morphine until pain free using a protocol (a bolus of 2mg morphine IV every ten minutes until pain free).

ELIGIBILITY:
Inclusion Criteria:

* women,
* 18years and older
* American Society of Anesthesiologists 1, 2,3,
* planned for radical mastectomy.

Exclusion Criteria:

* Neurological problems (central and peripheral)
* Bilateral mastectomy
* Body Mass Index > 33,
* Absolute contra-indication for ketorolac.
* Allergy/over-sensitiveness to levobupivacaine or local anesthetics of the same class
* Allergy/over-sensitiveness to dexmedetomidine or other alpha2 agonists (clonidine)
* Anatomic variations of the breast, pectoral region or axilla, noticed at clinical examination, including a pacemaker, Implantable Cardioverter Defibrillator, Port-a-Cath or other implantable device on the side that needs surgery.
* Participation in an other clinical trial within a period of four weeks before the beginning of this trial.
* Coagulopathy
* Infection or abcess in the region where the Block will be placed.
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-05-19 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Total postoperative opioid (morphine) consumption | 24 hours post procedure
  Milligrams of morphine used by the patient registrated by patient controlled intravenous analgesia delivery device (PCIA) during 24 hours after surgery

SECONDARY OUTCOMES:
Onset of postoperative pain | 24 hours post procedure
  Time between end of general anesthesia and a patients first demand of morphine registrated by PCIA.
Number of boluses morphine the patient asked for in the first 24 hours postoperative | 24 hours post procedure
  Amount of times the patient pushed the PCIA button even during lockout time period
Number of effectively delivered morphine boluses in the first 24 hours postoperatively | 24 hours post procedure
  Amount of times the patient pushed the PCIA button and morphine is delivered.

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Coppejans, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided